CLINICAL TRIAL: NCT03400397
Title: A Naturalistic Effectiveness Study of the Cool Kids Programme in Outpatient Psychiatric Clinics for Children in Southern Jutland, Denmark
Brief Title: An Effectiveness Study of the Cool Kids Programme
Status: Completed | Type: Observational
Sponsor: Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ida Drejer Djurhuus, Psychologist / clinical research assistent, Region of Southern Denmark
Other Study IDs: 16/37580
Record Dates: First submitted 2017-12-14; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Anxiety Disorder
Keywords: Anxiety; Child; Cognitive behaviour therapy; CBT; effectiveness; treatment; Cool Kids
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Treatment with the Cool Kids programme. The Cool Kids programme is a manualised cognitive behavioural treatment programme for children with anxiety disorders.
  Interventions: Other: Cool Kids programme

INTERVENTIONS:
Other: Cool Kids programme — A manualised cognitive behavioural treatment programme that consists of 10 session within 12-16 weeks each lasting 2 hours.

SUMMARY:
The aim of the present study is to investigate the effectiveness of the Cool Kids programme after implementation in two outpatient psychiatric clinics for children in Southern Jutland, Denmark. The Cool Kids programme is a manualised cognitive behavioural treatment programme for children aged 6 to 12 years with anxiety disorders. Previous efficacy studies have found that 60-80% of all children who complete the program show marked improvement. However, only one previous effectiveness study has ever been conducted. It is therefore relevant to examine whether the previously mentioned effect is maintained when the programme is implemented in a healthcare setting rather than a research setting.

DETAILED DESCRIPTION:
The study was conducted at two outpatient psychiatric clinics for children in Southern Jutland, Denmark.

Data was gathered from 55 patients who completed the Cool Kids programme as a treatment for anxiety disorder(s) from autumn 2013 to spring 2016. During the course of treatment both children and parents completed the Child Anxiety Life Interference Scale (CALIS) at baseline, post-treatment and at a 3-months follow-up booster-session. This data was originally gathered for internal quality assessment at the clinics. As the data was utilized for the present study in 2017, it has not been possible to control for confounding factors or influence the data-collection process.

All questionnaires were anonymised previous to being manually scored and keyed for secured electronic storage. Participants were excluded from the data analysis if they had one or more incomplete or missing CALIS. All statistical analysis was carried out in IBM SPSS 24 Statistical Software and consists of linear mixed effect models and one-way repeated measures ANOVAs.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnose: anxiety or obsessive-compulsive disorder according to ICD-10 criteria (F40-F42; F93)

Exclusion Criteria:

* comorbid diagnoses of:
* autism spectrum disorder
* conduct disorder
* untreated or severe ADHD
* low intelligence quotient (IQ)

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants had all been diagnosed with at least one anxiety or obsessive-compulsive disorder at the specialised child affective team at one of the two outpatient psychiatric clinics.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life and level of functioning measured by Child Anxiety Life Interference Scale (CALIS) | baseline, ended treatment (approx. 16-weeks) and 3-months follow-up
  Child Anxiety Life Interference Scale (CALIS) is a questionnaire that measures the degree of interference in level of functioning and quality of life caused by anxiety symptoms in 6- to 17-year-olds and their parents. CALIS is a scale for tracking treatment change.
  There are two versions of CALIS: a self-report questionnaire, and a parent-report questionnaire.
  All questions are answered on a 5-point Likert-scale with the choices: (0) Not at all, (1) Only a little, (2) Sometimes, (3) Quite a lot, and (4) A great deal. CALIS consists of 9 items in the self-report version and 16 items in the parent-report version split with respectively 9 and 7 items for interference in the child's and the parents' life. The self-report and parent-report scales for interference in the child's life is divided into two subscales: Outside Home (5 items) and At Home (4 items). The higher the score, the greater interference caused by anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ida M Djurhuus, MSc, Principal Investigator

IPD SHARING:
Plan to Share IPD: No